CLINICAL TRIAL: NCT01924962
Title: A Randomized Comparison of Recanalisation With Implantation of Cypher Sirolimus Eluting Coronary Stents and Medical Therapy
Brief Title: Recovery of Left Ventricular Function in Chronic Total Occluded Coronary Arteries
Acronym: REVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Responsible Party: Principal Investigator, Dr. Heinz Joachim Buettner, head of cath-lab department, University Heart Center Freiburg - Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK 1-2011
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Coronary Heart Disease
Keywords: chronic occlusion of coronary artery; left ventricular function; revascularisation
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- medical therapy (No Intervention): patients are treated with medical therapy only, intervention (stent) of other than (chronic occluded) target-vessel is allowed.
- revascularisation (Active Comparator): revascularisation and stent-implantation of chronic occluded coronary artery
  Interventions: Device: revascularisation

INTERVENTIONS:
Device: revascularisation — revascularisation of chronic occluded coronary artery
  Other Names: Cypher-stent
  Arms: revascularisation

SUMMARY:
The study is a randomised comparison of recanalisation of chronic occluded coronary arteries with implantation of Sirolimus eluting stents and medical therapy. Myocardial function and scar-size are determinated by using magnetic resonance imaging. The study hypothesis is the superiority of medical therapy over revascularisation.

DETAILED DESCRIPTION:
In the REVASC-study recovery of left ventricular function after recanalization of chronic total coronary occlusions (CTO) and implantation of sirolimus-eluting stents will be examined and compared to medical treatment. Extent of the scar, viable myocardium in the infarct zone and regional left ventricular function will be assessed by cardiac magnetic resonance. Patients with regional systolic left ventricular dysfunction of any degree in the supply territory of the CTO vessel will be randomized to either recanalization of the occluded coronary artery or to conservative therapy. It is of interest whether CTO patients will have an improvement in left ventricular function after late coronary reopening, regarding the high technical demands and costs of CTO recanalization.

ELIGIBILITY:
Inclusion Criteria:

* chronic total occlusion with thrombolysis in myocardial infarction (TIMI) 0 flow (or distal capillary reflow) of a native coronary artery with an estimated reference vessel diameter of 2.5 to 4.0 mm
* chronic total occlusion has more than 4 weeks duration
* the target vessel has not previously been treated with percutaneous coronary intervention
* the target vessel must be feasible for stent implantation
* patient has stable or unstable angina pectoris or a positive functional study for ischemia
* patient must be 18 years of age or older
* female subjects of childbearing age must have a negative pregnancy test within 7 days before procedure
* patient has been informed of the nature of the study and agrees to its
* provisions ans has written informed consent as approved by the Ethics Committee
* patient complies with all required post-procedure follow-up

Exclusion Criteria:

* a documented left ventricular function < 30%
* patient has a acute myocardial infarction (>3x normal creatine kinase (CK with presence of CK-MB) within 72 hours preceding the index procedure and CK has not returned to normal limits at the time of the procedure
* patients with known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, stainless steel or contrast media that cannot be adequately been pre-medicated
* patient has a platelet count of < 100000 cells/mm3 or > 700000 cells/m3, a white blood cell count of < 3000 cells/mm3 or documented or suspected liver disease
* patient has a history of bleeding diathesis or coagulopathy
* patient has suffered a cerebrovascular accident or transient ischemic attack within the past 6 months
* active peptic ulcer or upper gastrointestinal bleeding within the prior 6 months
* patients has a co-morbidity (i.e. cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, or is associated with limited life-expectancy (less than 2 years)
* the target vessel contains intraluminal thrombus
* the target vessel or lesson shows angiographic evidence of severe calcification
* patient has contraindications to magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2008-05-28 (Actual); Primary Completion 2016-08-14 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in regional left ventricular function at 9 months | 9 months
  Improvement of the left ventricular function in the territory of the chronically occluded coronary artery assessed by magnetic resonance imaging before revascularisation and at 9 months post-procedure. For regional left ventricular analysis, wall thickening and systolic inward motion will be determined in 12 segments in all short axis slices by the modified centerline method.

SECONDARY OUTCOMES:
Change from baseline in global left ventricular function at 6 months | 6 months
  Improvement of global left ventricular function (assessed by magnetic resonance imaging at baseline and 9 months post-procedure. For global left ventricular analysis, all short-axis slices from the apex to the base will be assessed. By planimetry of all short-axis views, left ventricular end-systolic volume (in milliliters), left ventricular end-diastolic volume (in milliliters), and ejection fraction (in percent) will be determined.
Changes from baseline in left ventricular volume at 6 months | 6 months
  Changes in diastolic and systolic volume indices (assessed by magnetic resonance imaging at baseline and 9 months post-procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Joachim Buettner, MD, Principal Investigator — Universitaets-Herzzentrum Freiburg-Bad Krozingen, Clinics for Cardiology and Angiology II, D-79189 Bad Krozingen, Germany
Locations (1):
- Universitäts Herzzentrum Freiburg Bad Krozingen, Bad Krozingen, Baden-Wurttemberg, Germany